CLINICAL TRIAL: NCT02710656
Title: Multicenter Randomized Controlled Trial Comparing Legflow - DCB (Cardionovum) Versus Bare Balloon Angioplasty for the Treatment of Atherosclerotic Disease in the Superficial Femoral & Popliteal Segment
Brief Title: Study Comparing Legflow Versus Bare Balloon Angioplasty for Treatment of Atherosclerotic Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardionovum GmbH (Industry)
Collaborators: Archer Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAGNIFICENT
Record Dates: First submitted 2016-03-07; First posted 2016-03-17 (Estimated); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Atherosclerosis
Keywords: Atherosclerosis; SFA; Poplitea; Drug coated balloon; Angioplasty; Restenosis; Peripheral artery disease (PAD)
MeSH Terms: conditions — Atherosclerosis; Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug Coated Balloon (DCB) - Legflow® (Experimental): Percutaneous balloon angioplasty performed with the investigational device, the paclitaxel eluting Legflow® balloon.
  Interventions: Device: Legflow® balloon
- Standard PTA - POBA (Active Comparator): Percutaneous balloon angioplasty performed with the clinical standard, that is, a non-drug eluting balloon (POBA, plain old balloon angioplasty).
  Interventions: Device: Standard PTA

INTERVENTIONS:
Device: Legflow® balloon — Percutaneous angioplasty performed with a Drug coated balloon (DCB) with Paclitaxel
  Other Names: Paclitaxel eluting balloon
  Arms: Drug Coated Balloon (DCB) - Legflow®
Device: Standard PTA — Percutaneous angioplasty performed with a standard balloon
  Other Names: POBA
  Arms: Standard PTA - POBA

SUMMARY:
A randomized multicentric study for endovascular treatment of patients with obstructive disease in the SFA (superficial femoral artery) and in the popliteal artery.

DETAILED DESCRIPTION:
This interventional study will collect data about the treatment of de novo lesions or restenotic lesions. Restenotic lesions that are previously DCB (drug coated balloon) treated or in-stent restenosis are excluded in this study.

The primary objective of this randomized study is to compare the efficacy of the DCB (Legflow - Cardionovum) versus POBA for the treatment of de novo lesions or restenosis in the SFA and in the popliteal artery (segment P1 -P2) by assessing the binary restenosis rate with duplex ultrasonography at 12 months.

The secondary endpoints are the assessment of the immediate procedural outcome, distribution of Rutherford, mortality, target lesion revascularization (TLR), target extremity revascularization (TER), amputation and anklebrachial index (ABI).

For each patient enrolled, data will be collected up to 12 months after the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must sign the informed consent form prior to the index-procedure.
2. Patient must be older than 18 years.
3. Patient with Rutherford 2, 3 and 4..
4. Target lesion is an occlusion or ≥70% stenosis (visual estimate) located in SFA or popliteal artery (P1 -P2).
5. Maximum length of the target lesion is 13 cm.
6. Target lesion is TASC A, B or C.
7. Target lesion is a de novo lesion or restenotic lesion (previously POBA treated, in-stent restenosis is not allowed).
8. Inflow arteries are free from hemodynamically significant obstruction (i.e. ≥ 50% diameter stenosis). It is allowed to treat inflow lesions during the index-procedure if the result is ≤ 30% diameter stenosis (treatment with DCB or DES is not allowed). Treatment of a non-target lesion in the target vessel is allowed if the nontarget lesion is considered to be an inflow lesion.
9. Popliteal artery P3 segment (below knee popliteal artery) is free from hemodynamically significant obstruction (i.e. ≥ 50%). Treatment of a lesion in this segment is not allowed during the index-procedure.
10. At least 1 patent (< 50% diameter stenosis) below-the-knee vessel (anterior tibial artery, posterior tibial artery or peroneal artery) till the ankle as confirmed by baseline angiography.

Exclusion Criteria:

1. Patient is already included in this study (recruitment of the contralateral leg is not allowed).
2. Patient has a known intolerance to antiplatelet therapy or contrast agent.
3. Patient with known sensitivity to Paclitaxel.
4. Patient is pregnant or patient intends to become pregnant within 1 year after the index-procedure.
5. Patient takes esomeprazole or omeprazole.
6. Patient with serum creatinine >2.0 mg/dL or renal dialysis.
7. Patient suffers from acute limb ischemia defined as any sudden decrease in limb perfusion causing a potential threat to limb viability.
8. Patient has a life expectancy <2 years.
9. Patient with Rutherford 0, 1 , 5 and 6.
10. Patient has a target lesion that is severely calcified (grade 3 and grade 4).
11. Patient with a TASC D lesion.
12. Patient has an acute thrombus or aneurysm in the target vessel.
13. Patient has a target lesion that cannot be crossed with a guidewire.
14. Target vessel has been treated previously with a DCB or a DES.
15. Treatment of outflow lesions during the index-procedure.
16. Patients with significant disease of all 3 infrapopliteal vessels (i.e. ≥ 50% diameter stenosis in each vessel).
17. Any scheduled surgery within 3 months after the index-procedure that would necessitate the discontinuation of clopidogrel.
18. Patients with previous bypass surgery involving the SFA.
19. Patient has cirrhosis of the liver.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Efficacy measured by binary restenosis rate | Until 12 months after procedure
  Binary restenosis rate determined by duplex ultrasonography at 1, 6 and 12 months afte procedure. Binary restenosis is defined as a re-obstruction ≥50% of the target lesion (peak systolic velocity ratio > 2.4).

SECONDARY OUTCOMES:
Immediate procedural outcome of percutaneous balloon angioplasty | From start of procedure surgery until completion of procedure surgery (Percutaneous balloon angioplasty)
  Investigator opinion of procedural and technical success of the percutaneous angioplasty. Opinion of investigator (yes/no) is recorded in the CRF for technical success and procedural success.
Rutherford | Baseline until 12 months after procedure
  Distribution of Rutherford stages during follow-up as compared to baseline.
Mortality | Until 12 months after procedure
  30-day mortality, 6-months mortality and overall mortality at 12 months.
Repeated target lesion revascularization (TLR) rate | Until 12 months after procedure
  TLR is defined as a repeated procedure (endovascular or surgical) due to a problem arising from the lesion (+1 cm proximally and distally to include edge phenomena) initially treated in surviving patients with preserved limb.
Repeated target extremity revascularization (TER) rate | Until 12 months after procedure
  TER is defined as a procedure (endovascular or surgical) due to a problem arising in the ipsilateral traject (iliac, femoropopliteal and below the knee arteries) remote from the lesion initially treated in surviving patients with preserved limb.
Minor and major amputation rate | Until 12 months after procedure
  Occurrence of minor (below the ankle) and major (above the ankle) amputations.
Ankle-Brachial Index (ABI) | Baseline until 12 months after procedure
  Reporting of Ankle-Brachial Index compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Peter Goverde, Dr., Principal Investigator — ZNA Stuivenberg
Locations (9):
- Belgium (5):
  - ZNA Stuivenberg, Antwerp
  - AZ Sint-Jan, Bruges
  - ZOL (Ziekenhuis Oost-Limburg), Genk
  - Jessa hospital, Hasselt
  - UZ Leuven, Leuven
- France (3):
  - CHU Bordeaux, Bordeau
  - CHU Cermont-Ferrand, Clermont-Ferrand
  - CH Mont-de-Marsan, Mont-de-Marsan
- Klinikum Arnsberg, Arnsberg, Germany

IPD SHARING:
Plan to Share IPD: No